CLINICAL TRIAL: NCT04991883
Title: Analysis of the Molecular Profile of the Mixofibrosarcoma of the Extremities: Diagnostic and Prognostic Impact
Brief Title: Analysis of the Molecular Profile of the Mixofibrosarcoma of the Extremities
Acronym: MFS
Status: Completed | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Other Study IDs: MFS
Record Dates: First submitted 2021-07-20; First posted 2021-08-05 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Sarcoma,Soft Tissue
Keywords: Mixofibrosarcoma
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: case series review of clinical and histological data — We will review all the medical records, radiological imaging, and histological data of these cases. The immunohistochemical analysis of the principal alterated genes identified in this tumor will be performed.

SUMMARY:
Single institution case series review with a histological diagnosis of mixofibrosarcoma of the extremities from 01 Jan 1993 to 01 Dec 2017.

The study will exam all the clinical, radiological, histological and immunohistochemical features of this tumour in all samples and in a limited serie of cases the presence of mutation of 50 genes cancer related.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients treated at Rizzoli Institute from 01 Jan 1993 to 01 Dec 2017
2. Diagnosis of mixofibrosarcoma of extremities
3. Histological slides/formalin-fixed paraffin-embedded tissue tumor (FFPE) blocks from archive available to perform the histology analysis and molecular analysis
4. Enough tumor biobanked material available for molecular analysis
5. Presence of the biobank signed informed consent
6. Written informed consent prior to any study-specific analysis and/or data collection

Exclusion Criteria:

1) Patients with histological diagnosis different from mixofibrosarcoma of extremities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of Mixofibrosarcoma treated at the Rizzoli Institute from 1 January 1993 up to 01 December 2017
Sampling Method: Probability Sample
Enrollment: 167 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
disease-free survival | at baseline (Day0)
  identify patients with different risk classes in terms of disease-free survival (local and systemic recurrence).
overall survival | at baseline (Day0)
  identify patients with different risk classes in terms of overall survival.

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mentzel T, Calonje E, Wadden C, Camplejohn RS, Beham A, Smith MA, Fletcher CD. Myxofibrosarcoma. Clinicopathologic analysis of 75 cases with emphasis on the low-grade variant. Am J Surg Pathol. 1996 Apr;20(4):391-405. doi: 10.1097/00000478-199604000-00001. PMID 8604805
- [Result] Gronchi A, Lo Vullo S, Colombo C, Collini P, Stacchiotti S, Mariani L, Fiore M, Casali PG. Extremity soft tissue sarcoma in a series of patients treated at a single institution: local control directly impacts survival. Ann Surg. 2010 Mar;251(3):506-11. doi: 10.1097/SLA.0b013e3181cf87fa. PMID 20130465
- [Result] Kaya M, Wada T, Nagoya S, Sasaki M, Matsumura T, Yamaguchi T, Hasegawa T, Yamashita T. MRI and histological evaluation of the infiltrative growth pattern of myxofibrosarcoma. Skeletal Radiol. 2008 Dec;37(12):1085-90. doi: 10.1007/s00256-008-0542-4. Epub 2008 Jul 16. PMID 18629459

DOCUMENTS (1):
  • Study Protocol (2020-06-12): https://cdn.clinicaltrials.gov/large-docs/83/NCT04991883/Prot_000.pdf